CLINICAL TRIAL: NCT06442787
Title: Analysis of Mandibular Proximal Segment Position Using Virtual Orthognathic Surgical Planning, Individualized Guides, and Osteosynthesis Plates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-54022451-050.04-150505
Record Dates: First submitted 2024-05-20; First posted 2024-06-04 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: CAD-CAM; Patients Specific Manufacturing; Osteotomy, Sagittal Split Ramus
Keywords: virtual surgical planning; orthognathic surgery; custom plate; mandibular condyle position

STUDY DESIGN:
Intervention Model Description: Orthognathic surgery is a surgical procedure performed to correct dentofacial deformities. In recent years, with the use of virtual surgical planning, cutting guides, and patient-specific osteosynthesis plates, highly predictable results can be achieved. While there are many positive reports regarding the use of patient-specific plates in maxillary positioning in orthognathic surgery, there is a lack of sufficient studies comparing the results obtained in mandibular positioning. Additionally, numerous designs of proximal segment positioning devices have been published, but comparative studies on their effectiveness have not been conducted. Therefore, a study comparing these approaches has been planned
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental): Orthognathic surgery will be performed (n=20) (control group)
  Interventions: Device: conventional splints
- group 2 (Active Comparator): Orthognathic surgery will be performed (n=20)
  Interventions: Device: cutting guides and positioning guides
- group 3 (Active Comparator): Orthognathic surgery will be performed (n=20)
  Interventions: Device: cutting guides and fixation plates

INTERVENTIONS:
Device: conventional splints — only intermediate and final splint will be used during the surgery
  Arms: control group
Device: cutting guides and positioning guides — patient's specific manufacturing cutting guide and positioning guide related with orthognathic surgery
  Arms: group 2
Device: cutting guides and fixation plates — patient's specific manufacturing cutting guide and fixation plates related with orthognathic surgery
  Arms: group 3

SUMMARY:
Orthognathic surgery is a surgical procedure performed to correct dentofacial deformities. In recent years, with the use of virtual surgical planning, cutting guides, and patient-specific osteosynthesis plates, highly predictable results can be achieved. While there are many positive reports regarding the use of patient-specific plates in maxillary positioning in orthognathic surgery, there is a lack of sufficient studies comparing the results obtained in mandibular positioning. Additionally, numerous designs of proximal segment positioning devices have been published, but comparative studies on their effectiveness have not been conducted. Therefore, a study comparing these approaches has been planned.

DETAILED DESCRIPTION:
Orthognathic surgery is a frequently used treatment method for correcting dentofacial deformities. Bilateral sagittal split osteotomy (BSSO), developed by Trauner and Obwegeser, is still used today with many design modifications. There is a potential for incorrect positioning of the proximal segment during fixation. Regarding mandibular setback surgery, many authors have reported a tendency for medial and posterior rotation of the proximal segment during the postoperative period. Proximal segment displacement may result from the condyle not seating properly in the fossa or from early contacts between the proximal and distal segments. These early contacts cause rotation of the proximal segment while the mandible is fixed. If the displacement exceeds the adaptive capacity of the condyle, a high rate of condylar resorption or postoperative relapse may occur. Various condylar positioning devices have been developed to overcome this issue.

The introduction of virtual surgical planning (VSP) has helped to overcome some of the errors and difficulties in model surgery and conventional surgical planning. Computer-aided design and manufacturing (CAD/CAM) splints have been shown to be accurate in transferring the surgical plan to real life, but some errors may still occur. Patient-specific 3D-printed osteosynthesis plates have been developed to overcome these errors. Many studies have reported high accuracy of these plates in the maxilla. However, some other studies have reported errors of 5-6 mm. Similar accuracy rates have been reported for the mandible, but there are fewer studies in this area.

VSP not only allows the surgeon to visualize 3D movements but also shows the osteotomy design, screw placement locations, fixation design, and early bone contacts. The amount of trimming of the distal segment is determined by examining whether any openings or narrowings occur after minor movements are made to the proximal segment based on the rotation of the distal segment or the complex "pitch" and "roll" movements of the occlusal plane. After all these movements are given with virtual planning, personalized cutting guides, positioning guides, and patient-specific plates are needed to transfer this plan to real life.

Recent developments in VSP have focused on accurately transferring preoperative planning to surgery. The most significant development in this regard is patient-specific plates and cutting guides. This technology enables surgeons and engineers to produce patient-specific cutting guides to determine the incision lines. These guides also determine the thickness of the bone in the areas where plate screws will be placed and ensure avoidance of tooth roots. Patient-specific plates are designed and manufactured to fit into pre-prepared holes and hold the osteotomized segments together in the desired position. Despite being a new technology, several studies have shown that VSP and patient-specific plates have better final surgical accuracies compared to VSP and splints.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals over 18 years of age
2. Patients with skeletal Class 2 and Class 3 malocclusion requiring bimaxillary orthognathic surgery
3. Patients who have undergone orthodontic treatment prior to surgery

Exclusion Criteria:

1. Patients with cleft lip and palate or craniofacial deformities
2. Oligodontia
3. Patients in whom the study protocol could not be continued due to intraoperative complications such as guide mismatch or bad split, or due to reasons such as inability to obtain postoperative CT scans
4. Patients with pre-existing temporomandibular joint disorders prior to surgery
5. Patients who have undergone previous orthognathic surgery
6. Patients with a history of maxillary or mandibular trauma
7. Patients requiring segmental maxillary surgery
8. Patients with bone metabolism disorders
9. Patients allergic to titanium
10. Pregnant individuals

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
mandibular condyle changes | in the first week after the surgery
  Firstly;
  The following reference planes and lines will be created on the Mimics (Materialise, Belgium, v21) software:
  * Frankfort Horizontal Plane (FHD): Right and left side porion and the plane passing through the right side orbitale
  * Midsagittal Reference Plane (MSR): Perpendicular to FHD, nasion and plane determined to pass through basion points Lateral Condylar Pole (LKK) (Right-Left): the outermost part of the condyle head point
  * Medial Condylar Pole (MKK) (Right-Left): innermost part of the condyle head point Linear and angular measurements to be made with these planes.

SECONDARY OUTCOMES:
Rate of the virtual surgical planning accuracy | in the first week after the surgery
  Postoperative CT data will be transferred to Mimics (Materialise, Belgium, v21) software in DICOM format. Here, a 3D head and jaw model will be obtained from this data. For this purpose, 24 cephalometric points will be selected in both models. In this software, an analysis containing these points will be created and the 2-dimensional linear distances between the preoperative and postoperative positions of these points will be calculated. The accuracy between preoperative and postoperative models will be evaluated in the Mimics software.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes